CLINICAL TRIAL: NCT02437747
Title: Local Drug Delivery of Aloe Vera Gel in Chronic Periodontitis Patients With Controlled Diabetes Mellitus
Brief Title: Locally Delivered Aloe Vera Gel in the Treatment of Chronic Periodontitis Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, Dr. Gurbani Kaur, Effect of locally delivered aloe vera gel as an adjunct to scaling and root planing in the treatment of chronic periodontitis patients with diabetes mellitus: Randomized controlled clinical trial, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPU/431(7) /2014
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus; Chronic Periodontitis
Keywords: clinical trial
MeSH Terms: conditions — Diabetes Mellitus; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRP+ Aloe Group (Experimental): Scaling and root planing was done along with application of aloe vera gel as an adjunct in selected sites.
  Interventions: Drug: SRP + Aloe
- SRP Group (Sham Comparator): Only scaling and root planing was done on the opposite side.
  Interventions: Procedure: SRP

INTERVENTIONS:
Drug: SRP + Aloe — Scaling and root planing along with aloe vera application was done
  Other Names: Korphad Ghar
  Arms: SRP+ Aloe Group
Procedure: SRP — Scaling and root planing was done
  Arms: SRP Group

SUMMARY:
A study on the effect of locally delivered aloe vera gel as an adjunct to scaling and root planing in the treatment of chronic periodontitis patients with controlled type II diabetes mellitus.The evaluation of Plaque Index, Gingival Index, Probing Pocket Depth, Relative Attachment Level at baseline, 6 weeks and 3 months and Glycosylated heamoglobin at baseline and 3 months.

DETAILED DESCRIPTION:
Aloe vera gel was locally delivered in the periodontal pockets of ≥ 5mm bilaterally in chronic periodontitis patients with diabetes under control.(HbA1c-6.6-8.6%).The study design had two groups-one in which scaling and root planing and local delivery of aloe vera gel and the other only scaling and root planing.

The evaluation of clinical parameters of PI, GI, PPD and RAL at baseline, 6 weeks and 3 months.

HbA1c evaluated at baseline and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 30 - 55 years from both genders.
2. Patients with controlled Type II Diabetes Mellitus (HbA1c < 7%) with Chronic periodontitis having ≥ 5mm periodontal pockets bilaterally atleast in one site.
3. Patients on oral hypoglycaemic agents.
4. Subjects who have not received periodontal therapy within preceding 6 months.
5. Patients willing to comply with all study related procedures.

Exclusion Criteria:

1. Subjects who have received antibiotic treatment in the preceding 3 months.
2. History of prolonged use of antibiotics/ steroids/ immunosuppressive agents /aspirin/ anticoagulants/ other medications including any other herbal products.
3. Pregnant or lactating women.
4. Smokers.
5. History of systemic diseases like hypertension, HIV, bone metabolic disorders, radiation therapy, Osteoporosis, immunosuppressive therapy, cancer etc.other than Diabetes.
6. Unwilling patients

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Clinical parameter of probing pocket depth | 3 months
  Clinically change in the probing pocket depth.

SECONDARY OUTCOMES:
Glycosylated haemoglobin | 3 months
  HbA1c levels evaluated at baseline and 3 months
Clinical parameter of plaque index | 3 months
  Change in the plaque index.
Clinical parameter of gingival index | 3 months
  Change in the gingival index.
Clinical parameter of relative attachment level | 3 months
  Change in the relative attachment level.

CONTACTS AND LOCATIONS:
Overall Officials: Archana Singh, MDS, Study Director — Dr.D.Y.Patil Vidyapeeth